CLINICAL TRIAL: NCT00967603
Title: Maintenance Therapy With Sunitinib or Observation in Metastatic Pancreatic Cancer: a Phase II Randomized Trial.
Brief Title: Maintenance Therapy With Sunitinib or Observation in Metastatic Pancreatic Cancer
Acronym: PACT-12
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Michele Reni, MD, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000643632; PACT-12 (Other: IRCCS San Raffaele); 2008-000814-65 (EudraCT Number)
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2009-12

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- observation (No Intervention): no therapy until progression
- sunitinib (Experimental): sunitinib until progression or for a maximum of 6 months
  Interventions: Drug: sunitinib

INTERVENTIONS:
Drug: sunitinib — oral sunitinib 37.5 mg daily
  Other Names: SUTENT
  Arms: sunitinib

SUMMARY:
RATIONALE: Sunitinib malate may stop the growth of tumor cells by blocking some of the tyrosine kinases needed for angiogenesis and cell growth. It is not yet known whether sunitinib malate is effective as maintenance therapy in delaying tumor progression in patients with metastatic pancreatic cancer who are progression-free after 6 months of induction chemotherapy.

PURPOSE: This randomized phase II trial is studying sunitinib malate as maintenance therapy to see how well it works compared with observation in avoiding tumor progression after induction chemotherapy in patients with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the 6-month progression-free survival of patients with metastatic pancreatic cancer without progression after 6 months of induction chemotherapy treated with sunitinib malate as maintenance therapy vs observation.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms:

* Arm I: Patients receive oral sunitinib malate once daily for up to 6 months in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients undergo observation only.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed metastatic pancreatic adenocarcinoma

  * Stage IV disease
* Received chemotherapy for a duration of 6 months
* No progressive disease for ≥ 6 months since beginning of induction chemotherapy (irrespective of regimen and response: stable disease, partial response, or complete response) demonstrated by the following:

  * Two consecutive CT or MR scans separated by ≥ 6 weeks
  * Normal or no CA19.9 increase > 20% during the last month

PATIENT CHARACTERISTICS:

* Karnofsky Performance Status 50-100%
* Adequate bone marrow, liver, and kidney function
* Normal thyroid gland function (euthyroid)
* Not pregnant or nursing
* No duodenal, gastric, or intestinal infiltration
* Able to take oral medication
* None of the following conditions related to cardiac disease, failure, or vascular disease including any of the following:

  * QTc interval prolongation
  * Congestive heart failure
  * Serious cardiac arrhythmias
  * Active coronary artery disease
  * Myocardial infarction
  * Ischemia
  * Cerebrovascular accident
  * Evidence of pre-existing uncontrolled hypertension
* No other malignancies except surgically cured carcinoma in situ of the cervix, basal or squamous cell carcinoma of the skin, or other adequately treated neoplasms for which the patient has been disease-free for ≥ 5 years

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No other prior chemotherapy apart from first-line treatment for pancreatic cancer
* More than 3 weeks and less than 8 weeks since prior chemotherapy (> 1 week in the case of fluorouracil as continuous infusion or capecitabine)
* No prior antiangiogenesis drugs, including any of the following:

  * Sunitinib malate
  * Sorafenib
  * Bevacizumab
  * AZD2171
  * Vatalanib
  * VEGF trap
  * Pazopanib
* More than 1 month since prior major surgical procedure and completely recovered
* More than 7-12 days since prior and no concurrent drugs that are known CYP3A4 inhibitors
* No concurrent drugs with potential anti-arrhythmic activity
* No concurrent thrombolytic agent at therapeutical dose
* No concurrent treatment with other experimental drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
6-month progression-free survival | every 2 months during therapy; every 3 months thereafter
  CT scan

SECONDARY OUTCOMES:
Response rate | every 2 months during therapy; every 3 months thereafter
  CT scan
Toxicity | monthly during therapy
  outpatient visit
OVERALL SURVIVAL | monthly
  outpatient visit
PROGRESSION-FREE SURVIVAL | every 2 months during therapy; every 3 months thereafter
  CT scan
endothelial circulating cells | baseline + every 2 months during therapy until progression
pharmacogenomics | baseline
pharmacokynetics | after 2 months of therapy
pharmacodynamics | baseline and every 2 months until progression

CONTACTS AND LOCATIONS:
Overall Officials: Michele Reni, MD, Principal Investigator — Istituto Scientifico H. San Raffaele
Locations (1):
- San Raffaele Scientific Institute, Milan, Italy